CLINICAL TRIAL: NCT04760483
Title: Soractelite(Tm) Transperineal Laser Ablation for Benign Prostatic Hyperplasia With Bladder Outlet Obstruction
Brief Title: Office Based Transperineal Laser Ablation for Benign Prostatic Hyperplasia HYPERPLASIA
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Urological Research Network, LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: URN-20201001
Record Dates: First submitted 2020-11-19; First posted 2021-02-18 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Male Urogenital Diseases; Genital Diseases, Male; Prostatic Disease; Prostatic Hyperplasia
Keywords: BPH; Prostate Enlargement; Bladder Outlet Obstruction
MeSH Terms: conditions — Male Urogenital Diseases; Genital Diseases, Male; Prostatic Diseases; Prostatic Hyperplasia; Urinary Bladder Neck Obstruction

STUDY DESIGN:
Intervention Model Description: Single arm study using intervention performed with Echolaser X4 that will be offered to men between 40 and 85 years of age, with moderate or severe international prostate symptoms scores and concomitant objective decrease in flow studies of at 30% consistent with bladder outlet obstruction
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Transperineal Laser Ablation for BPH (Experimental): Ceftriaxone 250 mg IM as antibiotic prophylaxis. Local Anesthesia: perineal skin will be infiltrated with 10 cc of Lidocaine 2% and then each neurovascular bundle will be infiltrated with 5 - 10 cc. Nitrous self-administered anesthesia will be available.
  One or two laser fibers from Echolaser x4 will be placed in each of the two prostate lobes using the plan. Treatment will be executed following Echolaser smart Interface planning, needles will follow targeted location using stepper grid under a transperineal approach in a sagittal plane. Ablation with 5 watts power per fiber, a total of ~ 1800 J will be delivered. We will evaluate pain measures and procedure tolerance using visual analog pain scale Upon completion we will measure coagulation zone with TRUS. Before discharge, trial of void will be conducted. Patients with a residual greater than 200 cc will have an indwelling catheter placed and will be discharged with it.
  Interventions: Device: SoracteLite(TM) TPLA for BPH

INTERVENTIONS:
Device: SoracteLite(TM) TPLA for BPH — see prior section
  Other Names: Laser ablation of prostate tissues

SUMMARY:
This study is set up as a phase I-II prospective, single center, interventional pilot study carried in Office setting under local anesthesia. It will assess the impact in quality of life and adverse events produced by transperineal laser ablation of the prostate (TPLA) in men 40 to 85 years of age with benign prostatic hypertrophy (BPH).

BPH is currently managed with medications (ie, alpha-1 adrenergic medications) and/or invasive approaches such as transurethral resection of prostate or surgical excision of prostate - robotic or open lead to relaxation or excision of the bladder neck. Such alteration of the bladder neck function or anatomy portends a significant and noticeable change on a male lifestyle, represented by absence of antegrade ejaculation among others. This study aims to evaluate the use of TPLA in the office setting under local anesthesia - greatly decreasing patient perioperative surgical risk. Moreover, it aims to determine safety profile and outcomes from TPLA therapy

The fundamental objective is to determine the feasibility and safety of TPLA in healthy men with LUTS due to BPH, successful performed in the outpatient office-based setting under local anesthesia. Secondary objectives include: 1-Uroflowmetry and Patient Reported Outcome Measures (PROMs) at three, six and 12 months; 2-Immediately spontaneous voiding post-TPLA; 3-Hematuria incidence after TPLA, measured by patient reporting; 4-LUTS after the treatment measured by IPSS; 5- Erectile function and presence of ejaculation after TPLA treatment and 6-Prostate volume changes using Transrectal ultrasound (TRUS) volume measurements

DETAILED DESCRIPTION:
INTRODUCTION

The Echolaser system (ELS - Elesta SpA. 50041, Calenzano (FI), Italy ), which consists of Echolaser X4 plus Echolaser Smart Interface is a new device for minimal invasive procedures. The system induces tissue coagulation thru a continuous 1064 nm laser wave. Light tissue interaction is reliable, reproducible, and safe. The laser fiber tip induces necrosis near the tip and coagulative effects deeper in tissues thru heat ablation. The body cleans up treated tissue over time. Much experience is gained with laser application in different organs. A preliminary study conducted in Europe by the investigators showed promising results (1)

About 4 out 5 men experience bothersome alterations in their voiding pattern. This pervasive condition usually begins in the 5th decade of life. These patients usually express complaints of Urinary urgency, frequency and nocturia as the sensation of incomplete voiding and decrease in the force of stream leading to stranguria. Lower Urinary Tract Symptoms (LUTS) is the common term that represents constellation of these symptoms, most triggered by prostate enlargement, commonly referred as Benign Prostatic Hyperplasia (BPH). Today management of BPH may call for medications such as alpha-blockers, 5 alpha reductase inhibitors, phosphodiesterase inhibitors or combination of them. In addition, there surgical approaches to improve BPH, they are based on cytodestruction or excision of prostate tissue. These surgical approaches range from office based minimally invasive to hospital based robotically conducted. Office based minimally invasive approaches are favored by patients given their low-risk nature, safety profile and avoidance of general or spinal anesthesia. Furthermore, minimally invasive approaches aim to preserve the bladder neck, this avoids alterations in sexual function such as retrograde ejaculation. Excision or resection of the bladder neck is a major step of definitive invasive approaches such as transurethral resection of prostate or surgical excision of prostate - robotic or open. Bladder neck resection portends a significant and noticeable change on a male lifestyle, represented by absence of antegrade ejaculation. This is a tradeoff that evokes hesitation in many men to resolve their BPH. Minimally invasive procedures have emerged aiming to relieve BPH without sacrificing the bladder neck. They carry two major advantages: preservation of ejaculation and absence of major anesthesia requirements, thus amenable to office setting execution. The latter provides significant saving to the health system and decreases post-operatory risks of adverse events in a not insignificant manner. The fundamental question raised to minimal invasive procedures relates to degree of subjective and objective response, durability of BPH relief, ability to wean off from medications and impact on quality of life, from a two domain - urinary and sexual perspective.

The ELS is a novel disruptive approach that allows a transperineal approach and provides for a safe and simultaneous multiple laser fiber energy delivery that translated in expediency and decreased procedure times. ELS has been safely conducted in men with BPH in the ambulatory setting, as a procedure called SoracteLiteTM transperineal laser ablation (TPLA), performed in men with LUTS due to BPH that were suboptimal candidates for surgery, they exhibited good tolerability with minimal adverse event profiles. To the investigators knowledge, there is no data or evaluation of its safety profile if/when conducted in an office setting under local anesthesia. Therefore, in this study the investigators aim to assess efficacy, tolerability, response and safety profile of SoracteLite™ TPLA conducted in men with LUTS due to BPH in the office setting.

Objective: The primary objective of this study is to assess efficacy, tolerability, short term response and safety profile of SoracteLite™ TPLA for LUTS due to BPH in healthy men. The secondary objectives are to evaluate quality of life changes in erectile and sexual function as the well as imaging volumetric changes in prostate size.

Study design: This study is set up as prospective, single center, interventional study.

Study population: The study will be offered to men ≥ 40 years of age, with moderate or severe international prostate symptoms scores and concomitant objective decrease in flow studies of at 30% consistent with bladder outlet obstruction (Qmax of 5 - 15 mL/sec, Elevated voiding pressures consistent with bladder outlet obstruction) Study Intervention Upon meeting inclusion and exclusion criteria, subjects will undergo prostate transperineal laser ablation planning and execution under local anesthesia using the ELS. Planning and execution will aim to destroy the prostate adenoma or transitional-anterior zones while sparing critical structures such as the urethra, neurovascular bundles, and bladder neck. The investigators anticipate between one and four laser fibers would be placed in the prostate to induce the laser coagulative necrosis required to achieve desired response.

Main study parameters/endpoints: Fundamental study parameters are efficacy and safety.

Efficacy will be measured in changes- improvement in IPSS score and uroflowmetry parameter as Qmax and Post void volume profile of the procedures measured by successfully completed SoracteLiteTM TPLA procedures. For safety, the main study parameter is the number of grade 3 or worse adverse events based on the CTCAE v5.0 within 30 days post procedure.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The risks for participation in this study are related to the SoracteLiteTM TPLA procedure. Laser fibers are introduced in the prostate by needles and these could injure and damage surrounding tissues. For example, plausibly, perforation of the urethra could lead to hematuria, clot retention and urinary tract infections. The laser energy delivery could damage vessels and nerves evoking erection changes, even loss. Thermal injuries from the laser could lead to communication with rectum leading to infections and fistulas. Furthermore, the prostatic tissue may become quite edematous triggering urinary retention that would require an indwelling catheter for several days or the weeks and may even trigger a need for of transurethral resection.

Granted, several precaution actions will be undertaken to reduce the patients' risk, such as:

1. Patients will be instructed to self-administer a fleet enema, the evening before and morning of the procedure.
2. The procedure will be performed under local anesthesia; thus, patient will be awake and able to provide feedback while it takes placed.
3. Single dose intravenous antibiotic prophylaxis with either cefuroxime or gentamicin will be provided.
4. Echolaser Smart Interface will be used for the planning of the treatment taking care of the safety distance in longitudinal and transversal US planes.
5. The laser fibers will be placed following the plan under live co-registered ultrasound guidance.
6. Laser ablation will be monitored in real time and restricted to the safety margins established on the plans, thus other critical anatomic areas will be spared.
7. Patients will be transferred to a recovery room and be discharge when subjectively they feel better and objectively have stable vital signs and full respiratory, cardiac, neurological and musculoskeletal capacities.

The following represent advantages of SoracteLiteTM TPLA: minimal invasive procedure; performance under local anesthesia; the intent is to treat transition-anterior zone, so called surgical capsule; urethral sparring, preservation of bladder neck and antegrade ejaculation, limited to absent need of indwelling catheterization.

The investigators aim to streamline the follow up following standard of care. Patients will be instructed to call if they perceive any adverse event. Patients will be contacted 30 days after procedure and an adverse event questionnaire will be administered. Subjective quality of life survey instruments will be administered 6 weeks and 3, 6 and 12 months from procedure date. Flow and volumetric studies will be conducted 3 months from procedure date.

In Conclusion, SoracteLiteTM TPLA will expose patients to intervention risks. However, is the investigators estimation and bias these will be favorable or equal to those observed with compared available standard minimal invasive treatment approaches. The burden is in our opinion acceptable.

ELIGIBILITY:
Inclusion Criteria:

* Presence of Lower Urinary Tract Symptoms (LUTS) measure by International Prostate Symptom Scores (IPSS) greater than 9
* Serum creatinine levels <1.5 ng/dl and GFR > 55
* Peak urinary flow rate (Qmax): ≥ 5 mL/sec to ≤ 15 mL/sec, with a minimum voided volume of ≥ 125 mL, measured with uroflowmetry, pressure flow studies or urodynamic investigation
* Post-void residual (PVR): ≤ 250 mL
* Prostate volume: ≥ 30 and ≤ 120 cc, measured by transrectal ultrasound
* Signed informed consent

Exclusion Criteria:

* Previous invasive prostate intervention (TURP, laser, ablation, etc.)
* History of prostate or bladder cancer
* Major neurological conditions such as Alzheimer's, Parkinson, Multiple sclerosis, ALS, spinal cord injury
* Evidence of neurogenic bladder
* Indwelling Foley catheter or clean intermittent catheterization (CIC) in the prior 30 days
* Inability or unwillingness to tolerate temporary discontinuation of anticoagulation or anti-platelet therapy
* Other conditions / status listed in full protocol

Ages: 40 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Males with prostates
Enrollment: 20 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2022-03-19 (Actual); Study Completion 2026-03-20 (Estimated)

PRIMARY OUTCOMES:
Feasibility and Tolerability of TPLA procedure | 30 minutes
  Treatment tolerance and satisfaction will be assessed using a visual analog pain scale during the procedure

SECONDARY OUTCOMES:
90 day Adverse Event profile of TPLA | 90 days
  Careful note of Emergent Adverse Events as assessed by CTCAE V5. Assessment will be upon removal of indwelling catheter, at the 15 day, 30 day and 90 day mark from the TPLA procedure date
Number of Participants with spontaneous voiding immediately following TPLA for BPH | 1 week
  Trial of void before patient is discharged. If fails a repeat voiding trial would be conducted within next 48 hours and if there is failure at 1 week.
Urinary Function following TPLA at the 3,6 & 12 months milestones | 12 months
  We will use standard validated questionnaires such as the international prostate symptoms score scale (I-PSS) as well as objective measures such as: urinary flow (average and max) and post void residuals at the identified milestones
Number of Participants having Erections and Ejaculation following TPLA at 3,6 & 12 months | 12 months
  Using SHIM scale min 1 max 25. Ability to have and sustain erections without any help or with help with a PDE5 inhibitor. Presence or absence of ejalucation

OTHER OUTCOMES:
Urinary Function and Sexual Function 2-3-4-5-years after procedure | 5 years
  We will use standard validated questionnaires such as the international prostate symptoms score scale (I-PSS) and Sexual Function inventory for Men (SHIM) during yearly in-person visit or via virtual interviews
Re-Treatment or Conversion to other surgical management | 5 years
  Will longitudinally observe the incidence of re-treatment with a similar procedure or conversion to other procedures such as: transurethral resection or ablation of the prostate, laser enucleation, REZUM, Urolift, Robotic open Open prostatectomy

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Bianco, MD, Principal Investigator — Urlogical Research Network
Locations (1):
- Urology Specialist Group, Hialeah, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Initial analysis after all subjects complete 3 month evaluation
Supporting Information: Study Protocol, SAP
Time Frame: 4 months after complete enrollment

REFERENCES:
- See also: Related Info — http://research.surgery